CLINICAL TRIAL: NCT02797860
Title: Comparison of Onset and Duration of Rocuronium Induced Neuromuscular Block Between 2nd Trimester Pregnant and Non-pregnant Women
Brief Title: Comparison of Onset and Duration of Rocuronium Between 2nd Trimester Pregnant and Non-pregnant Women
Status: Completed | Type: Observational
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Choi Eun MI, Hallym University Kangnam Sacred Heart Hospital, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: KangnamSHH
Record Dates: First submitted 2016-05-24; First posted 2016-06-14 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy
Keywords: Transabdominal cervicoisthmic cerclage; Rocuronium; Pregnant Women
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- transabdominal cervicoisthmic cerclage: Second Stage of Labor pregnant women who are scheduled for transabdominal cervicoisthmic cerclage due to incompetent internal os of cervix
  Interventions: Drug: Rocuronium
- control: women of childbearing age between 20 and 45
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — comparison of onset time and duration of rocuronium using Train of Four watch

SUMMARY:
Pregnancy is associated with major changes of the body's physiological status and composition.

These changes may modify the pharmacologic and/or pharmacokinetic profile of some drugs. Pharmacodynamic and pharmacokinetic changes in the 1st trimester during pregnancy are attributed to the following factors; Increase in plasma volume, heart rate and cardiac output; decrease in blood pressure due to decrease of systemic resistance and relative decrease of hepatic circulation and the aggravation of hepatic dysfunction. These changes intensify as pregnancy progresses into the 3rd trimester and take their effect on the onset time and duration of muscle relaxants.

Rocuronium and the steroidal non-depolarizing muscle relaxant like vecuronium is mostly excreted with bile by hepatic metabolism and classified as the FDA pregnancy category B, and is widely used in general anesthesia of pregnant women. Previous studies reported onset time of rocuronium is affected by cardiac output, blood circulation time of the whole body, and muscle perfusion. Accordingly, many researches were conducted under the assumption of onset time and duration being affected by physiologic changes during pregnancy. For example, in the research where vecuronium was used as muscle relaxant for pregnant woman undergoing C-sec, onset of vecuronium was significantly shorter than that of the control group and duration was longer. In a study investigating rocuronium used for patients right after delivery, onset time was shorter and duration was longer than that of the control group.

However, previous research mostly focused on the 3rd trimester, while there have been only a few studies of onset time and duration of rocuronium in non-obstetric surgery such as the transabdominal cervicoisthmic cerclage (TCIC) or Mcdonald surgery which are performed under general anesthesia during 2nd trimester. In this research, onset time and duration of rocuronium, which is widely used for general anesthesia in 2nd trimester pregnant females, will be compared with those of patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for Transabdominal cervicoisthmic cerclage under general anesthesia or patients scheduled for elective open abdominal surgery.
* The American Society of Anesthesiologists physical status class one or two
* female between 20 and 45

Exclusion Criteria:

* Patients with liver disease
* Patients with kidney disease
* Patients with Diabetes mellitus or heart disease
* Patients with asthma or Bronchial hypersensitivity
* Patients with a drug allergy
* Patients BMI under 18.5 or over 27

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients scheduled for Transabdominal cervicoisthmic cerclage under general anesthesia
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
onset time of rocuronium | until T1 of Train of Four watch is suppressed to 0%,assessed up to 5 minutes

SECONDARY OUTCOMES:
duration of rocuronium | until T1 of Train of Four watch is recovered to 25%,assessed up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Eun Mi Choi, MD, Study Director — Hallym University Kangnam Sacred Heart Hospital
Locations (1):
- Kangnam sacred heart hospital, Seoul, Yeongdeungpo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robson SC, Hunter S, Boys RJ, Dunlop W. Serial study of factors influencing changes in cardiac output during human pregnancy. Am J Physiol. 1989 Apr;256(4 Pt 2):H1060-5. doi: 10.1152/ajpheart.1989.256.4.H1060. PMID 2705548
- [Result] Capeless EL, Clapp JF. When do cardiovascular parameters return to their preconception values? Am J Obstet Gynecol. 1991 Oct;165(4 Pt 1):883-6. doi: 10.1016/0002-9378(91)90432-q. PMID 1951547
- [Result] Greiss FC Jr, Anderson SG. Effect of ovarian hormones on the uterine vascular bed. Am J Obstet Gynecol. 1970 Jul 15;107(6):829-36. doi: 10.1016/s0002-9378(16)34033-9. No abstract available. PMID 5429013
- [Result] Chapman AB, Abraham WT, Zamudio S, Coffin C, Merouani A, Young D, Johnson A, Osorio F, Goldberg C, Moore LG, Dahms T, Schrier RW. Temporal relationships between hormonal and hemodynamic changes in early human pregnancy. Kidney Int. 1998 Dec;54(6):2056-63. doi: 10.1046/j.1523-1755.1998.00217.x. PMID 9853271
- [Result] Bernstein IM, Ziegler W, Badger GJ. Plasma volume expansion in early pregnancy. Obstet Gynecol. 2001 May;97(5 Pt 1):669-72. doi: 10.1016/s0029-7844(00)01222-9. PMID 11339913
- [Result] Van Thiel DH, Gavaler JS. Pregnancy-associated sex steroids and their effects on the liver. Semin Liver Dis. 1987 Feb;7(1):1-7. doi: 10.1055/s-2008-1040558. No abstract available. PMID 3589711
- [Result] Esbjorner E, Jarnerot G, Sandstrom B, Ostling G. Serum albumin reserve for bilirubin binding during pregnancy in healthy women. Obstet Gynecol. 1989 Jan;73(1):93-6. PMID 2909046
- [Result] Wierda JM, Kleef UW, Lambalk LM, Kloppenburg WD, Agoston S. The pharmacodynamics and pharmacokinetics of Org 9426, a new non-depolarizing neuromuscular blocking agent, in patients anaesthetized with nitrous oxide, halothane and fentanyl. Can J Anaesth. 1991 May;38(4 Pt 1):430-5. doi: 10.1007/BF03007578. PMID 1829656
- [Result] Munoz HR, Gonzalez AG, Dagnino JA, Gonzalez JA, Perez AE. The effect of ephedrine on the onset time of rocuronium. Anesth Analg. 1997 Aug;85(2):437-40. doi: 10.1097/00000539-199708000-00034. No abstract available. PMID 9249127
- [Result] Szmuk P, Ezri T, Chelly JE, Katz J. The onset time of rocuronium is slowed by esmolol and accelerated by ephedrine. Anesth Analg. 2000 May;90(5):1217-9. doi: 10.1097/00000539-200005000-00041. PMID 10781483
- [Result] Hans P, Brichant JF, Hubert B, Dewandre PY, Lamy M. Influence of induction of anaesthesia on intubating conditions one minute after rocuronium administration: comparison of ketamine and thiopentone. Anaesthesia. 1999 Mar;54(3):276-9. doi: 10.1046/j.1365-2044.1999.00703.x. PMID 10364866
- [Result] Baraka A, Jabbour S, Tabboush Z, Sibai A, Bijjani A, Karam K. Onset of vecuronium neuromuscular block is more rapid in patients undergoing caesarean section. Can J Anaesth. 1992 Feb;39(2):135-8. doi: 10.1007/BF03008643. PMID 1347489
- [Result] Camp CE, Tessem J, Adenwala J, Joyce TH 3rd. Vecuronium and prolonged neuromuscular blockade in postpartum patients. Anesthesiology. 1987 Dec;67(6):1006-8. doi: 10.1097/00000542-198712000-00028. No abstract available. PMID 2891326
- [Result] Sakurai Y, Uchida M, Aiba J, Mimura F, Yamaguchi M, Kakumoto M. [Effects of pregnancy on the onset time of rocuronium]. Masui. 2014 Mar;63(3):324-7. Japanese. PMID 24724444
- [Result] Puhringer FK, Sparr HJ, Mitterschiffthaler G, Agoston S, Benzer A. Extended duration of action of rocuronium in postpartum patients. Anesth Analg. 1997 Feb;84(2):352-4. doi: 10.1097/00000539-199702000-00020. PMID 9024027